CLINICAL TRIAL: NCT03870971
Title: User Evaluation of the Invasive Component of the CNOGA TensorTip COMBO GLUCOMETER (CoG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciema UG (Other)
Collaborators: Cnoga Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CNG-NGM-005
Record Dates: First submitted 2019-02-12; First posted 2019-03-12 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Blood Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood glucose measurement — After the patient has performed the manual reading, the investigator or staff member will obtain another capillary blood sample and a reference reading by means of the YSI 2300 Stat plus analyzer will be performed and recorded. If patients need more than one attempt to get a successful blood glucose reading, the number of attempts will be documented. A questionnaire needs to filled by the participant

SUMMARY:
Open label, prospective, comparative, multi-center study. All participants will get an introduction to the invasive component of the TENSORTIP COG by means of the instructions for use in English language only (incl. an illustrated short manual) and will be asked to perform a reading without further device training. Thereafter, a healthcare professional will perform an additional reading with the reference method (YSI 2300 STAT plus). In addition, blood will be drawn for determination of hematocrit. In the study, a minimum of 10 test strip vials that cover a minimum of 3 strip lots will be used. In addition multiple devices will be employed. After completion of the study the study participants will be given a questionnaire to fill out.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 1 or type 2 diabetes or healthy
* Subjects who are able to complete informed consent form (by him/herself or by his/her guardian);
* 18 years old and above;

Exclusion Criteria:

* Does not meet inclusion criteria;
* Subjects with any other severe disease in the discretion of the investigator
* Not capable to read English user instructions at the discretion of the patient
* Pregnancy or Nursing mothers
* Any condition that may prevent participants from successful participation in the trial (in discretion of the investigator)
* Illiteracy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
measurement performance | up to 1 day
  invasive CoG (study device) blood glucose measurement in comparison to blood glucose measurment of a comparator device (YSI 2300 STAT Plus).

CONTACTS AND LOCATIONS:
Locations (1):
- Rainier Clinical Research Center, Inc., Renton, Washington, United States

IPD SHARING:
Plan to Share IPD: No